CLINICAL TRIAL: NCT06903520
Title: Clinical Correlation Study Between Anomalous Pancreaticobiliary Ductal Junction and Malignant Tumors of the Biliary System and the Establishment of an AI-based Automated Recognition System
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lu Wenping, director, Chinese PLA General Hospital
Other Study IDs: 2023-037-01
Record Dates: First submitted 2025-03-28; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pancreaticobiliary Maljunction
MeSH Terms: conditions — Pancreaticobiliary Maljunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the occurrence of pancreaticobiliary maljunction (PBM) in the Chinese population, the characteristics of various subtypes, and the relationship between PBM and malignant tumors of the biliary system. To explore the general clinical characteristics of patients with mild bile duct dilation but who have not been clinically diagnosed with choledochal cysts, as well as the relationship between these characteristics and malignant tumors of the biliary system. To develop and evaluate a deep learning method for machine learning of Magnetic resonance cholangiopancreatography (MRCP) images, enabling fully automated detection of pancreaticobiliary maljunction.

ELIGIBILITY:
Inclusion Criteria:

Cases that were hospitalized and underwent Magnetic resonance cholangiopancreatography (MRCP) examination at the First Medical Center of Chinese People's Liberation Army General Hospital.

Exclusion Criteria:

1. Patients aged less than 18 years old;
2. Those with unclear diagnosis;
3. Cases with missing or poor-quality imaging data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with pancreaticobiliary maljunction
Sampling Method: Non-Probability Sample
Enrollment: 2439 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The incidence rate of malignant tumors of the biliary system | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, China